CLINICAL TRIAL: NCT06237309
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of a Single Dose of REGN5381, an NPR1 Monoclonal Antibody Agonist, in Patients With Chronic Heart Failure With Reduced Ejection Fraction
Brief Title: REGN5381 in Adult Participants With Heart Failure With Reduced Ejection Fraction
Acronym: NATRIX-BNP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R5381-HF-22118; 2023-508568-31-00 (EU CTIS Number)
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Heart failure with reduced ejection fraction (HFrEF); Reduced ejection fraction; N-terminal pro-brain natriuretic peptide (NT-proBNP) hormone
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part A1 High Dose (Experimental): Single ascending dose cohort
  Interventions: Drug: REGN5381
- Part A1 Low Dose (Experimental): Single ascending dose cohort
  Interventions: Drug: REGN5381
- Part A1 Optional (Experimental): Single ascending dose cohort
  Interventions: Drug: REGN5381
- Part A2 High Dose, sacubitril-valsartan group (Experimental): Single ascending dose cohort
  Interventions: Drug: REGN5381
- Part A2 Low Dose, sacubitril-valsartan group (Experimental): Single ascending dose cohort
  Interventions: Drug: REGN5381
- Placebo for Part A2, sacubitril-valsartan group (Placebo Comparator)
  Interventions: Drug: Placebo
- Part A2 High Dose, Low estimated glomerular filtration rate (eGFR) group (Experimental): Single ascending dose cohort. Note: This group has been closed
  Interventions: Drug: REGN5381
- Part A2 Low Dose, Low eGFR group (Experimental): Single ascending dose cohort. Note: This group has been closed
  Interventions: Drug: REGN5381
- Placebo for Part A2, Low eGFR group (Placebo Comparator): Note: This group has been closed
  Interventions: Drug: Placebo
- Part B High Dose (Experimental)
  Interventions: Drug: REGN5381
- Part B Low Dose (Experimental)
  Interventions: Drug: REGN5381
- Part A1 and Part B Placebo Only (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN5381 — Single dose intravenous (IV) infusion
  Arms: Part A1 High Dose; Part A1 Low Dose; Part A1 Optional; Part A2 High Dose, Low estimated glomerular filtration rate (eGFR) group; Part A2 High Dose, sacubitril-valsartan group; Part A2 Low Dose, Low eGFR group; Part A2 Low Dose, sacubitril-valsartan group; Part B High Dose; Part B Low Dose
Drug: Placebo — Single dose IV infusion
  Arms: Part A1 and Part B Placebo Only; Placebo for Part A2, Low eGFR group; Placebo for Part A2, sacubitril-valsartan group

SUMMARY:
This study is researching an experimental drug called REGN5381 (called "study drug"). The study is focused on patients with heart failure with reduced ejection fraction (ie, the heart is not functioning as well as it should).

The aim of the study is to see how safe, tolerable, and effective the study drug is.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the study drug less effective or could lead to side effects)

DETAILED DESCRIPTION:
Enrollment for the Part A2 low eGFR cohort has been closed

ELIGIBILITY:
Key Inclusion Criteria

1. Body mass index (BMI) between 18 and 45 kg/m^2, inclusive, at initial screening visit
2. Diagnosis of chronic heart failure
3. Left ventricular ejection fraction 20-49% by echocardiogram performed within 3 months of screening
4. Plasma NT-proBNP ≥800 pg/mL (or ≥1000 pg/mL if in atrial fibrillation) at screening (visit 1) and NT-proBNP ≥600 pg/mL (or ≥800 pg/mL if in atrial fibrillation) approximately 30 days prior to randomization (visit 5)
5. Receiving optimized standard of care therapy for heart failure as described in the protocol
6. Sacubitril-valsartan treatment:

   a. Treatment with sacubitril-valsartan at screening and at baseline permitted in Part A2 sacubitril-valsartan cohort and in Part B if supported by safety data from the Part A2 sacubitril-valsartan cohort as described in the protocol
7. Estimated Glomerular Filtration Rate (eGFR) levels:

   1. eGFR of ≥30 mL/min/1.73 m2 according to locally used formula (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] preferred), at screening (visit 1) or approximately 30 days prior to randomization (visit 5) as described in the protocol

Key Exclusion Criteria

1. Hospital discharge within 180 days of anticipated randomization
2. Resting SBP that remains out of range after two repeated measurements prior to randomization as described in the protocol
3. Current or recent diagnosis of acute coronary syndrome or myocardial infarction as described in the protocol
4. History of symptomatic autonomic dysfunction as evidenced by orthostatic hypotension and/or syncope
5. Unexplained syncope <12 months prior to initial screening or during the Run-in period
6. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disease, as assessed by the investigator that may confer unreasonable risk to the participant's participation in the study
7. Uncorrected congenital heart disease
8. Cardiac surgery within 6 months prior to screening or any planned surgery during the study
9. Implantation of a cardiac resynchronization therapy device in the prior 90 days, or planned during the study, or planned device optimization 30 days prior to randomization or during the study
10. Current chronic lung disease requiring long-term oxygen therapy

Note: Other protocol-defined inclusion/ exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in circulating N-Terminal pro-Brain Natriuretic Peptide (NTproBNP) | Day 8

SECONDARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Events (TEAEs) | Through week 16
Severity of TEAEs | Through week 16
Change from baseline in circulating NT-proBNP | Week 2
Change from baseline in circulating NT-proBNP | Week 3
Change from baseline in circulating NT-proBNP | Week 4
Change from baseline in circulating NT-proBNP | Up to week 16
Change from baseline in Systolic Blood Pressure (SBP) | Each visit through week 16
Change from baseline in Diastolic Blood Pressure (DBP) | Each visit through week 16
Change from baseline in Mean Arterial Pressure (MAP) | Each visit through week 16
Change from baseline in Heart Rate (HR) | Each visit through week 16
Concentrations of REGN5381 in serum | Through week 16
Incidence of Anti-Drug Antibodies (ADAs) to REGN5381 | Through week 16
Magnitude of ADAs to REGN5381 | Through week 16

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Administrator, Study Director — Regeneron Pharmaceuticals
Locations (44):
- United States (4):
  - Arensia Exploratory Medicine Clinic, Phoenix, Arizona
  - Harbor UCLA Medical Center, Torrance, California
  - Flourish Research - Miami (Kendall) (Formerly Clinical Site Partners), Miami, Florida
  - Flourish Research - Orlando (Formerly Clinical Site Partners), Winter Park, Florida
- Belgium (8):
  - Grand Hopital de Charleroi, Gilly, Hainaut
  - Anima Research Center, Alken, Limburg
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams Brabant
  - Algemeen Ziekenhuis St Jan Brugge Oostende Av, Bruges, West Flanders
  - Algemeen Ziekenhuis Groeninge, Kortrijk, West Vlaanderen
  - AZ Oostende, Ostend, West Vlaanderen
  - Centre Hospitalier Regional de la Citadelle, Liège
- Bulgaria (3):
  - MHAT Haskovo, Haskovo
  - University Multiprofile Hospital for Active Treatment Plovdiv, Plovdiv
  - Arensia Exploratory Medicine Clinic at MBAL Sveta Sofia, Sofia
- Czechia (4):
  - Fakultni Nemocnice v Motole, Prague, Central Bohemian
  - University Hospital Brno, Brno, South Moravian
  - Medicus Services s.r.o., Brandýs nad Labem-Stará Boleslav
  - Edumed, Jaroměř
- Arensia Exploratory Medicine at the Research Institute of Clinical Medicine, Tbilisi, Georgia
- Greece (4):
  - First Cardiology Clinic University of Athens, Athens, Attica
  - Athens Naval Hospital, Athens, Attikh
  - General University Hospital Attikon, Chaïdári
  - Larissa University Hospital, Larissa
- Pmsi Republican Clinical Hospital Timofei Mosneaga, Chisinau, Moldova
- Poland (5):
  - Wojewodzki Szpital Zespolony - Ludwik Rydygier Provincial Hospital, Torun, Kuyavian-Pomeranian Voivodeship
  - UCK Medical University of Warsaw, Warsaw, Masovian Voivodeship
  - Medical University of Lodz, Lodz
  - NZOZ Gemini, Żychlin
  - Clinmedica Research sp zo.o., Skierniewice, Łódź Voivodeship
- Romania (2):
  - Arensia Exploratory Medicine Clinic at Monza Bucharest, Bucharest
  - Sc Arensia Exploratory Medicine Srl, Cluj-Napoca
- South Africa (4):
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - Into Research, Groenkloof, Gauteng
  - Dr M I Sarvan,R Moodley & partners, Durban, KwaZulu-Natal
  - Kuils River Hospital, Kuils River, Western Cape
- South Korea (4):
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Severance Hospital at Yonsei University College of Medicine, Seoul, Seodaemun-gu
  - Korea University Guro Hospital, Seoul
- Spain (4):
  - Virgen de las Montañas Hospital, Villamartín, Cadiz
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Virgen Macarena Unidad Coronaria 1 planta, Seville
  - Hospital Arnau de Vilanova, Valencia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/